CLINICAL TRIAL: NCT00005279
Title: Tucson Epidemiology Study of Chronic Obstructive Lung Diseases
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 2000; P50HL014136 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2002-05

CONDITIONS: Asthma; Bronchitis; Emphysema; Lung Diseases, Obstructive; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Asthma; Bronchitis; Emphysema; Lung Diseases, Obstructive; Pulmonary Disease, Chronic Obstructive

SUMMARY:
To determine the natural history, etiology, and interrelationships of emphysema, chronic bronchitis, asthma, and related airways obstructive diseases. Also, to determine the relationship of acute lower respiratory tract illnesses in infants and children to the development of subsequent chronic lung disorders.

DETAILED DESCRIPTION:
BACKGROUND:

The Tucson Epidemiology Study of Chronic Obstructive Lung Diseases had been supported by the Specialized Center of Research (SCOR) mechanism since 1971. The SCOR mechanism was instituted to advance basic knowledge and to generate the most effective techniques and methods of clinical management and prevention.

In 1970, the chronic obstructive lung diseases (COLD) of bronchitis, emphysema, and asthma were the tenth leading cause of death in the United States. At that time United States mortality from emphysema had been increasing at the rate of 20-25 percent per year. In 1969 the death rate for COLD as a whole was 15.6 per 100,000 and that rate was considered to be only about one-half of all those deaths in which COLD was either an underlying or an important contributory cause. By 1986 COLD had risen to be the fifth leading cause of death in the United States with a death rate of 31.3 per 100,000.

By 1972 many prevalence surveys had been conducted in the United States and abroad on specific subgroups of populations. At that time, most longitudinal studies were limited in the scope of examinations conducted, dealt with restricted age groups, and conducted few studies of familial concordance of diseases. The Tucson study was designed to include a wide age span, family units, and a variety of features relating to reversible or irreversible obstructive lung disease.

Studies have provided evidence relating acute lower respiratory tract illnesses in the first few years of life to the development of chronic lung disease in later life. Epidemiologic studies have demonstrated that geographic areas with high morbidity and mortality rates due to chronic obstructive lung disease among adults are also likely to show a high incidence of respiratory illness among children. A number of risk factors may be associated with lower respiratory tract illness in children. Some studies suggested that familial or genetic factors may predispose certain children to respiratory disorders early in life. Family size, viral and bacterial infections, allergic reaction, air pollution, gas stoves, formaldehyde, and passive smoking have all been implicated. Research was needed on the interrelationships of potential risk factors and lower respiratory tract infections in producing chronic respiratory disease.

DESIGN NARRATIVE:

The Tucson Study of Chronic Obstructive Lung Diseases was longitudinal in design. By 1986, nine surveys had been completed on 70 percent of the same population surveyed at baseline in 1972. Data collected in the surveys included basic standardized questionnaires and maximum expiratory flow volume (MEFV) curves using the same pneumotachograph equipment. Additional questionnaires were included on smoking, medical and occupational history, socio-economic characteristics, and height and weight measurements. Blood was sampled for studies of alpha-1-antitrypsin level. Several surveys included allergy skin testing, blood pressure, and anthropometric measurements. Studies of the 504 out-migrants continued since 1982. Twelve surveys were planned to insure a follow-up of at least 15 years on all adults.

Funding represented approximately 26 percent of the dollars of the Specialized Center of Research in Chronic Diseases of the Airways (P5OHL14136) used to support the Tucson Study.

Childrens' Respiratory Study of Tucson was also longitudinal in design and assessed the role of infectious, physiologic, immunologic, allergic, genetic, environmental, and familial factors in the development of acute and chronic lower respiratory tract illnesses in childhood. Enrollment of the study population and their families occurred between May 1980 and October 1984. Healthy infants were enrolled within a few days of birth, at which time baseline data were collected. Cord and 9-month bloods were evaluated for a number of immunologic tests. In the first few months of life, prior to any lower respiratory tract illnesses, a subset of the population underwent pulmonary function testing. During lower respiratory tract illness, specimens were obtained for viral, chlamydial, and mycoplasma cultures and tests. Environmental factors evaluated included passive smoking, number of siblings, overcrowding, and air pollution. Data collection was continued on the children and their family members over the years.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1971-06; Study Completion 1997-11 (Actual)

REFERENCES:
- [Background] Burrows B (Ed): Chronic Respiratory Disease, Med Clin North Am, W.B. Saunders Co, May 1973
- [Background] Burrows B. Editorial: Early detection of airways obstruction. Chest. 1974 Mar;65(3):239-40. doi: 10.1016/s0012-3692(15)36309-1. No abstract available. PMID 4813828
- [Background] Lebowitz MD, Burrows B. Air pollution and respiratory illness. Ariz Med. 1973 Aug;38(8):543-7. No abstract available. PMID 4581576
- [Background] Knudson RJ, Burrows B. Early detection of obstructive lung diseases. Med Clin North Am. 1973 May;57(3):681-90. doi: 10.1016/s0025-7125(16)32267-2. No abstract available. PMID 4573465
- [Background] Nelson DC, Burrows B, Knudson RJ. A device for recording flow and volume data in population surveys. J Appl Physiol. 1973 Aug;35(2):304-6. doi: 10.1152/jappl.1973.35.2.304. No abstract available. PMID 4723041
- [Background] Morse JO, Lebowitz MD, Knudson RJ, Burrows B. A community study of the relation of alpha1-antitrypsin levels to obstructive lung diseases. N Engl J Med. 1975 Feb 6;292(6):278-81. doi: 10.1056/NEJM197502062920602. PMID 1078596
- [Background] Diener CF, Burrows B. Further observations on the course and prognosis of chronic obstructive lung disease. Am Rev Respir Dis. 1975 Jun;111(6):719-24. doi: 10.1164/arrd.1975.111.6.719. PMID 1137239
- [Background] Burrows B: Prognosis of the Bronchial and Emphysematous Types. In: Chron Obstr Lung, Stuttgart: Schattauer, pp. 171-173, 1975
- [Background] Lebowitz MD, Knudson RJ, Burrows B. Tucson epidemiologic study of obstructive lung diseases. I: Methodology and prevalence of disease. Am J Epidemiol. 1975 Aug;102(2):137-52. doi: 10.1093/oxfordjournals.aje.a112141. PMID 1155443
- [Background] Lebowitz MD, Burrows B. Tucson epidemiologic study of obstructive lung diseases. II: Effects of in-migration factors on the prevalence of obstructive lung diseases. Am J Epidemiol. 1975 Aug;102(2):153-63. doi: 10.1093/oxfordjournals.aje.a112142. PMID 1155444
- [Background] Lebowitz M, Burrows B: The Relationship of Acute Respiratory Illness History as a Precursor of Chronic Obstructive Lung Disease. (Abs) in Proc. Soc. Epidem. Res., Am J Epidemiol, 100:511, 1974
- [Background] Lebowitz MD, Morse JO, Knudson RJ, Barbee R, Burrows B. Respiratory disorders in Tucson: preliminary observations. Ariz Med. 1975 Apr;32(4):329-31. No abstract available. PMID 1078974
- [Background] Burrows B, Lebowitz MD. Characteristics of chronic bronchitis in a warm, dry region. Am Rev Respir Dis. 1975 Sep;112(3):365-70. doi: 10.1164/arrd.1975.112.3.365. PMID 1163892
- [Background] Lebowitz MD, Burrows B. Respiratory symptoms related to smoking habits of family adults. Chest. 1976 Jan;69(1):48-50. doi: 10.1378/chest.69.1.48. PMID 1244287
- [Background] Lebowitz M: Aerosol Usage and Respiratory Symptomatology. Arch Environ Health. (Presented at Food and Drug Administration Hearings, Washington, D.C, Dec. 16-18, 1974
- [Background] Barbee RA, Lebowitz MD, Thompson HC, Burrows B. Immediate skin-test reactivity in a general population sample. Ann Intern Med. 1976 Feb;84(2):129-33. doi: 10.7326/0003-4819-84-2-129. PMID 766679
- [Background] Burrows B, Lebowitz MD, Barbee RA. Respiratory disorders and allergy skin-test reactions. Ann Intern Med. 1976 Feb;84(2):134-9. doi: 10.7326/0003-4819-84-2-134. PMID 1252041
- [Background] Barbee R, Lebowitz MD, Morse JO, Burrows B: The Relationships of Atopy and Smoking Habits to Respiratory Disease in a General Population. (Abs) J Clin Res, 24:121A, 1976
- [Background] Knudson RJ, Slatin RC, Lebowitz MD, Burrows B. The maximal expiratory flow-volume curve. Normal standards, variability, and effects of age. Am Rev Respir Dis. 1976 May;113(5):587-600. doi: 10.1164/arrd.1976.113.5.587. PMID 1267262
- [Background] Knudson RJ, Burrows B, Lebowitz MD. The maximal expiratory flow-volume curve: its use in the detection of ventilatory abnormalities in a population study. Am Rev Respir Dis. 1976 Nov;114(5):871-9. doi: 10.1164/arrd.1976.114.5.871. PMID 791036
- [Background] Lebowitz MD, Burrows B. Comparison of questionnaires: the BMRC and NHLI respiratory questionnaires and a new self-completion questionnaire. Am Rev Respir Dis. 1976 May;113(5):627-35. doi: 10.1164/arrd.1976.113.5.627. PMID 1267264
- [Background] Lebowitz MD. Aerosol usage and respiratory symptoms. Arch Environ Health. 1976 Mar-Apr;31(2):83-6. doi: 10.1080/00039896.1976.10667195. PMID 1259474
- [Background] Taussig L, Lebowitz MD: Cough and Wheeze Syndromes in Children. (abs) Am Rev Respir Dis, 113 (part 2):45, 1976
- [Background] Burrows B, Knudson RJ, Cline MG, Lebowitz MD. Quantitative relationships between cigarette smoking and ventilatory function. Am Rev Respir Dis. 1977 Feb;115(2):195-205. doi: 10.1164/arrd.1977.115.2.195. PMID 842934
- [Background] Burrows B, Knudson RJ, Lebowitz MD. The relationship of childhood respiratory illness to adult obstructive airway disease. Am Rev Respir Dis. 1977 May;115(5):751-60. doi: 10.1164/arrd.1977.115.5.751. PMID 857715
- [Background] Burrows B, Lebowitz MD, Knudson RJ. Epidemiologic evidence that childhood problems predispose to airways disease in the adult (an association between adult and pediatric respiratory disorders). Pediatr Res. 1977 Mar;11(3 Pt 2):218-20. No abstract available. PMID 846771
- [Background] Knudson RJ, Lebowitz MD, Burton AP, Knudson DE. The closing volume test: evaluation of nitrogen and bolus methods in a random population. Am Rev Respir Dis. 1977 Mar;115(3):423-34. doi: 10.1164/arrd.1977.115.3.423. PMID 842954
- [Background] Knudson RJ, Lebowiz MD. Comparison of flow-volume and closing volume variables in a random population. Am Rev Respir Dis. 1977 Dec;116(6):1039-45. doi: 10.1164/arrd.1977.116.6.1039. PMID 931180
- [Background] Lebowitz MD. Smoking habits and changes in smoking habits as they relate to chronic conditions and respiratory symptoms. Am J Epidemiol. 1977 Jun;105(6):534-43. doi: 10.1093/oxfordjournals.aje.a112417. PMID 868857
- [Background] Lebowitz MD. Occupational exposures in relation to symptomatology and lung function in a community population. Environ Res. 1977 Aug;14(1):59-67. doi: 10.1016/0013-9351(77)90066-4. No abstract available. PMID 891505
- [Background] Lebowitz MD: A Critical Examination of Factorial Ecology and Social Area Analysis for Epidemiological Research. J Az Acad Sci, 12:86-90, 1977
- [Background] Lebowitz MD. The relationship of socio-environmental factors to the prevalence of obstructive lung diseases and other chronic conditions. J Chronic Dis. 1977 Sep;30(9):599-611. doi: 10.1016/0021-9681(77)90058-3. No abstract available. PMID 903391
- [Background] Lebowitz MD, Burrows B. Quantitative relationships between cigarette smoking and chronic productive cough. Int J Epidemiol. 1977 Jun;6(2):107-13. doi: 10.1093/ije/6.2.107. PMID 892975
- [Background] Lebowitz MD, Burrows B. The relationship of acute respiratory illness history to the prevalence and incidence of obstructive lung disorders. Am J Epidemiol. 1977 Jun;105(6):544-54. doi: 10.1093/oxfordjournals.aje.a112418. PMID 868858
- [Background] Lebowitz MD, Johnson WM, Kaltenborn W: Coccidioidin Skin Test Reactivity and Cross-Reactivity with Histoplasmin in a Tucson Population. Coccidioidomycosis (Ajello, L, Ed.) Selected Papers from 3rd Intr. Coccidioidomycosis Symposium, Tucson, Az., Nov, 1976, Miami, Fla.: Symposia Specialists 1977
- [Background] Morse JO, Lebowitz MD, Knudson RJ, Burrows B. Relation of protease inhibitor phenotypes to obstructive lung diseases in a community. N Engl J Med. 1977 May 26;296(21):1190-4. doi: 10.1056/NEJM197705262962102. PMID 300842
- [Background] Lebowitz MD: Alcohol Consumption, Smoking and Respiratory Symptomatology. (abs) Am J Epidemiol, 106:248, 1977 (Presented at the 10th Annual Meeting Soc. Epidemiol Res., Seattle, June 16, 1977
- [Background] Lebowitz MD, Knudson RJ, Armet D, Kaltenborn W, Burrows B: Longitudinal Changes in Lung Function and Respiratory Symptoms. (abs) IEA Proc, 1977, 193 (Presented at the 8th Scientific Meeting of IEA, San Juan, Puerto Rico September 1977
- [Background] Morse JO, Lebowitz MD, Knudson RJ: Value of Antitrypsin Screening. (Correspondence) N Engl J Med, 297:454-455, 1977
- [Background] Lebowitz MD: Temporal Analysis of Acute Respiratory Symptoms, Aero-Allergens and Air Pollution. (abs) IEA Proc., 194 (Presented at the 8th Scientific Meeting of IEA, San Juan, Puerto Rico, September 1977
- [Background] Burrows B: Course and Prognosis in Advanced Disease. In: Chronic Obstructive Pulmonary Disease, Petty T (Ed), New York: Marcel Dekker, Inc., Chapter 2, pp. 23-33, 1978
- [Background] Burrows B. [Approaches to the prevention and management of chronic nonspecific respiratory diseases]. Bull Int Union Tuberc. 1978 Dec;53(4):327-35. No abstract available. French. PMID 756310
- [Background] Dodge RR, Reed CE, Barbee RA. The absence of a relationship between serum precipitins and pulmonary disease in a community. Chest. 1978 May;73(5):608-12. doi: 10.1378/chest.73.5.608. PMID 648212
- [Background] Lebowitz MD, Knudson RJ, Morse JO, Armet D. Closing volume and flow volume abnormalities in alpha(1)-antitrypsin phenotype groups in a community population. Am Rev Respir Dis. 1978 Jan;117(1):179-81. doi: 10.1164/arrd.1978.117.1.179. PMID 304327
- [Background] Lorber DB, Kaltenborn W, Burrows B. Responses to isoproterenol in a general population sample. Am Rev Respir Dis. 1978 Nov;118(5):855-61. doi: 10.1164/arrd.1978.118.5.855. PMID 736356
- [Background] Morse JO. alpha1-antitrypsin deficiency (first of two parts). N Engl J Med. 1978 Nov 9;299(19):1045-8. doi: 10.1056/NEJM197811092991905. No abstract available. PMID 360063
- [Background] Knudson RJ, Lebowitz MD. Maximal mid-expiratory flow (FEF25-75%): normal limits and assessment of sensitivity. Am Rev Respir Dis. 1978 Mar;117(3):609-10. doi: 10.1164/arrd.1978.117.3.609. No abstract available. PMID 629492
- [Background] Kerrebijn KF, Neijens HJ. Comparison of flow-volume and closing volume variables in a random population. Am Rev Respir Dis. 1978 Aug;118(2):445. doi: 10.1164/arrd.1978.118.2.445. No abstract available. PMID 697193
- [Background] Barbee RA, Lebowitz MD, Ryan KJ, Tennican P. Coccidioidomycosis: Alias San Joaquin Valley fever. Med Times. 1979 Apr;107(4):2D (20)-4D (20), 8D (20), 15D (20). No abstract available. PMID 431348
- [Background] Brown WG, Halonen MJ, Kaltenborn WT, Barbee RA. The relationship of respiratory allergy, skin test reactivity, and serum IgE in a community population sample. J Allergy Clin Immunol. 1979 May;63(5):328-35. doi: 10.1016/0091-6749(79)90127-1. No abstract available. PMID 429712
- [Background] Knudson RJ, Lebowitz MD, Slatin RC. The timing of the forced vital capacity. Am Rev Respir Dis. 1979 Feb;119(2):315-8. doi: 10.1164/arrd.1979.119.2.315. PMID 434602
- [Background] Loughlin GM, Taussig LM. Pulmonary function in children with a history of laryngotracheobronchitis. J Pediatr. 1979 Mar;94(3):365-9. doi: 10.1016/s0022-3476(79)80572-7. PMID 423015
- [Background] McDonagh DJ, Nathan SP, Knudson RJ, Lebowitz MD. Assessment of alpha-1-antitrypsin deficiency heterozygosity as a risk factor in the etiology of emphysema. Physiological comparison of adult normal and heterozygous protease inhibitor phenotype subjects from a random population. J Clin Invest. 1979 Feb;63(2):299-309. doi: 10.1172/JCI109303. PMID 311786
- [Background] Nathan SP, Lebowitz MD, Knudson RJ. Spirometric testing. Number of tests required and selection of data. Chest. 1979 Oct;76(4):384-8. doi: 10.1378/chest.76.4.384. PMID 477423
- [Background] Traver GA, Cline MG, Burrows B. Predictors of mortality in chronic obstructive pulmonary disease. A 15-year follow-up study. Am Rev Respir Dis. 1979 Jun;119(6):895-902. doi: 10.1164/arrd.1979.119.6.895. PMID 453709
- [Background] Burrows B. Course and prognosis of patients with chronic airways obstruction. Chest. 1980 Feb;77(2 Suppl):250-1. doi: 10.1378/chest.77.2_supplement.250. No abstract available. PMID 7357895
- [Background] Knudson RJ, Armet DB, Lebowitz MD. Reevaluation of tests of small airways function. Chest. 1980 Feb;77(2 Suppl):284-6. doi: 10.1378/chest.77.2.284. No abstract available. PMID 7357909
- [Background] Garfield M, Sugihara S, Abraham TA, Lebowitz MD, Burrows B: Characteristics of Individuals With Rapidly Declining FEV1 Identified Within a General Population. (abs) Am Rev Respir Dis, 121(#4, part 2):138, 1980. Presented at the ATS Annual Meeting, Washington, D.C., May 21, 1980
- [Background] Abraham TA, Garfield M, Sugihara S, Lebowitz MD, Burrows B: Methacholine Inhalation Challenge in Normal Individuals Using the Maximum and Partial Flow Curves With an Assessment of Diurnal Variation. (abst) Am Rev Respir Dis, 121 (#4, Part 2):53, 1980
- [Background] Helsing KJ, Comstock GW, Speizer FE, Ferris BG, Lebowitz MD, Tockman MS, Burrows B. Comparison of three standardized questionnaires on respiratory symptoms. Am Rev Respir Dis. 1979 Dec;120(6):1221-31. doi: 10.1164/arrd.1979.120.6.1221. No abstract available. PMID 517854
- [Background] Burrows B, Hasan FM, Barbee RA, Halonen M, Lebowitz MD. Epidemiologic observations on eosinophilia and its relation to respiratory disorders. Am Rev Respir Dis. 1980 Nov;122(5):709-19. doi: 10.1164/arrd.1980.122.5.709. PMID 7447155
- [Background] Dodge RR, Burrows B. The prevalence and incidence of asthma and asthma-like symptoms in a general population sample. Am Rev Respir Dis. 1980 Oct;122(4):567-75. doi: 10.1164/arrd.1980.122.4.567. PMID 7436122
- [Background] Burrows B: Prognostic Factors in Chronic Obstructive Pulmonary Disease. Pract Cardiol, 6(10):61-69, 1980
- [Background] Wagener JS, Taussig LM, Burrows B, Hernried L, Boat T: Comparison of Lung Function and Survival Patterns Between Cystic Fibrosis and Emphysema or Chronic Bronchitis Patients. Perspectives in Cystic Fibrosis, Proceedings of the 8th International Cystic Fibrosis Congress, Toronto, May 1980
- [Background] Turner-Warwick M, Burrows B, Johnson A. Cryptogenic fibrosing alveolitis: clinical features and their influence on survival. Thorax. 1980 Mar;35(3):171-80. doi: 10.1136/thx.35.3.171. PMID 7385089
- [Background] Burrows B, Taussig LM. "As the twig is bent, the tree inclines" (perhaps). Am Rev Respir Dis. 1980 Dec;122(6):813-6. doi: 10.1164/arrd.1980.122.6.813. No abstract available. PMID 7458055
- [Background] Turner-Warwick M, Lebowitz M, Burrows B, Johnson A. Cryptogenic fibrosing alveolitis and lung cancer. Thorax. 1980 Jul;35(7):496-9. doi: 10.1136/thx.35.7.496. PMID 7434310
- [Background] Turner-Warwick M, Burrows B, Johnson A. Cryptogenic fibrosing alveolitis: response to corticosteroid treatment and its effect on survival. Thorax. 1980 Aug;35(8):593-9. doi: 10.1136/thx.35.8.593. PMID 7444826
- [Background] Lebowitz MD. Respiratory indicators. Environ Res. 1981 Jun;25(1):225-35. doi: 10.1016/0013-9351(81)90091-8. No abstract available. PMID 7238465
- [Background] Burrows B, Halonen M, Barbee RA, Lebowitz MD. The relationship of serum immunoglobulin E to cigarette smoking. Am Rev Respir Dis. 1981 Nov;124(5):523-5. doi: 10.1164/arrd.1981.124.5.523. PMID 7305105
- [Background] Barbee RA, Halonen M, Lebowitz M, Burrows B. Distribution of IgE in a community population sample: correlations with age, sex, and allergen skin test reactivity. J Allergy Clin Immunol. 1981 Aug;68(2):106-11. doi: 10.1016/0091-6749(81)90167-6. PMID 7251998
- [Background] Lebowitz MD. Epidemiological recognition of occupational pulmonary diseases. Clin Chest Med. 1981 Sep;2(3):305-16. No abstract available. PMID 7028383
- [Background] Lebowitz MD. Respiratory symptoms and disease related to alcohol consumption. Am Rev Respir Dis. 1981 Jan;123(1):16-9. doi: 10.1164/arrd.1981.123.1.16. PMID 7458081
- [Background] Frank R, Lebowitz MD: The Risk of Staying In. (Editorial) Am Rev Respir Dis, 124:522, 1981
- [Background] Lebowitz MD. The relationship among silica, silicosis, and lung carcinoma. Ariz Med. 1981 Aug;38(8):596-8. No abstract available. PMID 6268025
- [Background] Burrows B. An overview of obstructive lung diseases. Med Clin North Am. 1981 May;65(3):455-71. doi: 10.1016/s0025-7125(16)31509-7. No abstract available. PMID 7242173
- [Background] Barbee RA, Brown WG, Kaltenborn W, Halonen M. Allergen skin-test reactivity in a community population sample: correlation with age, histamine skin reactions and total serum immunoglobulin E. J Allergy Clin Immunol. 1981 Jul;68(1):15-9. doi: 10.1016/0091-6749(81)90117-2. PMID 7240595
- [Background] Lebowitz MD, Thompson HC, Strunk RC. Subjective psychological symptoms in outpatient asthmatic adolescents. J Behav Med. 1981 Dec;4(4):439-49. doi: 10.1007/BF00846152. PMID 7338897
- [Background] Landau LI, Taussig LM, Burrows B, Cline M, Lebowitz MD, Knudson R: Sex Differences in Growth Velocity of Lung Function Assessed From Longitudinal Measurements in Healthy Subjects Age 6 to 25 Years. Australian Ped J, 17(2):145, 1981
- [Background] Dodge R, Burrows B: Chronic Bronchitis and Emphysema. In: Prognosis Contemporary Outcomes of Disease. (JF Fries, GE Ehrlich, Eds) Bowie, MD: Charles Press Publishers, pp. 228-231, 1981
- [Background] Burrows B. Pulmonary disease. Postgrad Med. 1981 Apr;69(4):100-1. doi: 10.1080/00325481.1981.11715733. No abstract available. PMID 27452826
- [Background] Burrows B: Management of Chronic Obstructive Lung Disease. Drug Ther, pp. 127-133, Nov. 1981
- [Background] Halonen M, Barbee RA, Lebowitz MD, Burrows B. An epidemiologic study of interrelationships of total serum immunoglobulin E, allergy skin-test reactivity, and eosinophilia. J Allergy Clin Immunol. 1982 Feb;69(2):221-8. doi: 10.1016/0091-6749(82)90103-8. No abstract available. PMID 7056953
- [Background] Coaker L, Lebowitz MD, Abraham T, Garfield M, Suqihara S, Burrows B: Methacholine Challenge: The Correlation of Smoking With Airway Response in Symptomatic and Asymptomatic Subjects. Am Rev Respir Dis, 125(#4, part 2):253, 1982
- [Background] Lebowitz MD, Knudson RJ, Robertson G, Burrows B. Significance of intraindividual changes in maximum expiratory flow volume and peak expiratory flow measurements. Chest. 1982 May;81(5):566-70. doi: 10.1378/chest.81.5.566. PMID 7075275
- [Background] Lebowitz MD, Knudson RJ, Armet D, Kaltenborn W, Burrows B: Smoking and Longitudinal Changes in Lung Function and Respiratory Symptoms. Indian J Chest Dis, Special Number: Smoking and Health, pp. 47-56, 1982
- [Background] Burrows B: Irreversible Airways Obstruction and Asthma. Pract Cardiol, 8(7):69-81, 1982
- [Background] Offord KP, Gleich GJ, Barbee RA, Dunnette SL, Miller RD. Serum IgD in subjects with and without chronic obstructive pulmonary disease: a previous finding restudied. Am Rev Respir Dis. 1982 Jul;126(1):118-20. doi: 10.1164/arrd.1982.126.1.118. PMID 7091896
- [Background] Burrows B, Halonen M, Lebowitz MD, Knudson RJ, Barbee RA. The relationship of serum immunoglobulin E, allergy skin tests, and smoking to respiratory disorders. J Allergy Clin Immunol. 1982 Sep;70(3):199-204. doi: 10.1016/0091-6749(82)90042-2. PMID 7108071
- [Background] Lebowitz MD. Multivariate analysis of smoking and other risk factors for obstructive lung diseases and related symptoms. J Chronic Dis. 1982;35(9):751-8. doi: 10.1016/0021-9681(82)90099-6. PMID 7107807
- [Background] Lebowitz MD, Armet DB, Knudson RJ: The Effect of Passive Smoking on Pulmonary Function in Children. Environ Internat'l, 8:371-374, 1982
- [Background] Lebowitz MD: The Effects of Alcohol Ingestion on the Lung. Pract Cardiol, 8:101-104, 1982
- [Background] Lebowitz M, O'Rourke M, Dodge R, Holberg C, Corman G, Hoshaw R, Pinnas J, Barbee R, Sneller M: The Adverse Health Effects of Biological Aerosols, Other Aerosols, and Microclimate Indoors on Asthmatics and Non-Asthmatics. Environ Internat'l, 8:375-380, 1982
- [Background] Burrows B: The Natural History of Airflow Limitation. Med Clin North Am, pp. 2157-2162, April 1982
- [Background] Burrows B: The Natural History of Airflow Limitation. Med Internat'l, 1:955-956, 1982
- [Background] Lebowitz MD, Dodge R, Holberg C: The Effects of the Environment on Pulmonary Function in Children, In: Proceedings of the National Congress on Pediatric Bronchopneumonology. D. Castello (Ed), Turin: Italian Ped. Bronchopneumonal. Assn., 1982
- [Background] Bloom, JW, Sugihara S, Garfield M, Abraham T, Knudson RJ: Factors Associated With Rapid Decline in Lung Function. Am Rev Respir Dis, 125:258S, 1982
- [Background] Knudson RJ, Lebowitz MD, Holberg CJ, Burrows B. Changes in the normal maximal expiratory flow-volume curve with growth and aging. Am Rev Respir Dis. 1983 Jun;127(6):725-34. doi: 10.1164/arrd.1983.127.6.725. PMID 6859656
- [Background] Lebowitz MD. Health effects of indoor pollutants. Annu Rev Public Health. 1983;4:203-21. doi: 10.1146/annurev.pu.04.050183.001223. No abstract available. PMID 6860438
- [Background] Lebowitz MD. The effects of pressurized aerosols on respiratory symptoms and physiology. Sci Total Environ. 1983 Jul;29(1-2):19-27. doi: 10.1016/0048-9697(83)90031-1. PMID 6612325
- [Background] Burrows B. A clinical trial of efficacy of antiproteolytic therapy: can it be done? Am Rev Respir Dis. 1983 Feb;127(2):S42-3. doi: 10.1164/arrd.1983.127.2P2.S42. No abstract available. PMID 6600891
- [Background] Bloom J, Sugihara S, Garfield M, Abraham T, Knudson RJ: Characteristics of Individuals With Accelerated Declines in Lung Function. Chest, 85(6):18S-19S, 1983
- [Background] Burrows B, Lebowitz MD, Barbee RA, Knudson RJ, Halonen M. Interactions of smoking and immunologic factors in relation to airways obstruction. Chest. 1983 Dec;84(6):657-61. doi: 10.1378/chest.84.6.657. PMID 6641298
- [Background] Lebovitz MD. [Temporary changes in acute respiratory symptoms depending on allergens and atmospheric air pollution]. Przegl Lek. 1983;40(11):777-82. No abstract available. Polish. PMID 6669730
- [Background] Toxic substances in the atmospheric environment. Critical review discussion papers. J Air Pollut Control Assoc. 1983 Sep;33(9):827-43. doi: 10.1080/00022470.1983.10465648. No abstract available. PMID 6630750
- [Background] Lebowitz MD, Dodge RR, Holberg CJ, Corman G, Boyer B: Daily Symptoms Related to Indoor Pollution in Adult Asthmatics and Non-Asthmatics. Am J Epidemiol, 118(3):419, 1983
- [Background] Buist AS, Burrows B, Eriksson S, Mittman C, Wu M. The natural history of air-flow obstruction in PiZ emphysema. Report of an NHLBI workshop. Am Rev Respir Dis. 1983 Feb;127(2):S43-5. doi: 10.1164/arrd.1983.127.2P2.S43. No abstract available. PMID 6600892
- [Background] Burrows B: COPD: A New Look at DX and RX of an Old Problem. Modern Med, pp. 114-126, March, 1983
- [Background] Burrows B, Knudson RJ, Quan SF, Kettel LJ: Respiratory Disorders: A Pathophysiologic Approach, 2nd Ed. Revised. Chicago: Year Book Medical Publishers, Inc. 1983
- [Background] Burrows B: Early Diagnosis of COPD: Value of Annual Spirometric Examination of Smokers. Pract Cardiol, 9:143-150, 1983
- [Background] Burrows B: Trends in Respiratory Medicine. Todays Therapeutic Trends, 1:11-20, 1983
- [Background] Sobonya RE, Burrows B. The epidemiology of emphysema. Clin Chest Med. 1983 Sep;4(3):351-8. No abstract available. PMID 6357599
- [Background] Burrows B, Cline MG, Knudson RJ, Taussig LM, Lebowitz MD. A descriptive analysis of the growth and decline of the FVC and FEV1. Chest. 1983 May;83(5):717-24. doi: 10.1378/chest.83.5.717. PMID 6839813
- [Background] Lebowitz MD: Potential Respiratory Problems Within the Home Environment, In: Energy, Air Pollution and Health: Seminar Proceedings. W. Linn (Ed) New York: American Lung Association, pp. 76-87, 1983
- [Background] Lebowitz MD, Waller RE, Jacobsen M, Kostrezewski J, Hasegawa Y (Eds): Guidelines on Studies in Environmental Epidemiology. (Environmental Health Criteria 27) Geneva: World Health Organization, 1983
- [Background] Lebowitz MD, et al: Organization and Conduct of Studies. Chapter 5 in: Lebowitz MD, Waller RE, Jacobsen M, Kostrezewski J, Hasegawa Y, (Eds) Guidelines on Studies in Environmental Epidemiology. (Environmental Health Criteria 27) Geneva: World Health Organization, pp. 211-261, 1983
- [Background] Bloom JW, Farland AM, Halonen M, Burrows B: Pneumococcus Specific IgE in Cigarette Smokers. Am Rev Respir Dis, 129(4):A191, 1984
- [Background] Lebowitz MD, Knudson R, Burrows B: Risk Factors for Airway Obstructive Diseases: A Multiple Logistics Approach. Chest, 85(6):11S-12S, 1984
- [Background] Lebowitz MD, Knudson RJ, Burrows B. Family aggregation of pulmonary function measurements. Am Rev Respir Dis. 1984 Jan;129(1):8-11. doi: 10.1164/arrd.1984.129.1.8. PMID 6703487
- [Background] Lebowitz MD, Barbee R, Burrows B. Family concordance of IgE, atopy, and disease. J Allergy Clin Immunol. 1984 Feb;73(2):259-64. doi: 10.1016/s0091-6749(84)80017-2. PMID 6699309
- [Background] Bloom JW, Kaltenborn WT, Paoletti P, Camilli A, Lebowitz MD. Respiratory effects of non-tobacco cigarettes. Br Med J (Clin Res Ed). 1987 Dec 12;295(6612):1516-8. doi: 10.1136/bmj.295.6612.1516. PMID 3122882
- [Background] Knudson RJ, Bloom JW, Kaltenborn WT, Burrows B, Lebowitz MD. Assessment of air vs helium-oxygen flow-volume curves as an epidemiologic screening test. Chest. 1984 Sep;86(3):419-23. doi: 10.1378/chest.86.3.419. PMID 6468002
- [Background] Knudson RJ, Bloom JW, Knudson DE, Kaltenborn WT. Subclinical effects of smoking. Physiologic comparison of healthy middle-aged smokers and nonsmokers and interrelationships of lung function measurements. Chest. 1984 Jul;86(1):20-9. doi: 10.1378/chest.86.1.20. PMID 6734286
- [Background] Lebowitz MD. The effects of environmental tobacco smoke exposure and gas stoves on daily peak flow rates in asthmatic and non-asthmatic families. Eur J Respir Dis Suppl. 1984;133:90-7. No abstract available. PMID 6586467
- [Background] Robertson G, Lebowitz MD. Analysis of relationships between symptoms and environmental factors over time. Environ Res. 1984 Feb;33(1):130-43. doi: 10.1016/0013-9351(84)90014-8. PMID 6692807
- [Background] Bloom JW, Burrows B: Diseases Associated With Airflow Limitation, In: Current Pulmonology, Vol. 5 (Simmons DH, Ed) John Wiley & Sons, Inc., pp. 255-281, 1984
- [Background] Burrows B: Possible Pathogenetic Mechanisms in Chronic Airflow Obstruction. Chest, 85S:13S-15S, 1984
- [Background] Bruce RM, Cohen BH, Diamond EL, Fallat RJ, Knudson RJ, Lebowitz MD, Mittman C, Patterson CD, Tockman MS. Collaborative study to assess risk of lung disease in Pi MZ phenotype subjects. Am Rev Respir Dis. 1984 Sep;130(3):386-90. doi: 10.1164/arrd.1984.130.3.386. PMID 6332562
- [Background] Camilli A, Paoletti P, Lebowitz MD: Types of Occupational Exposures, Respiratory Symptoms and Lung Function. Am Rev Respir Dis, 129 (#4, part 2):A170, 1984
- [Background] Higgins MW, Keller JB, Landis JR, Beaty TH, Burrows B, Demets D, Diem JE, Higgins IT, Lakatos E, Lebowitz MD, et al. Risk of chronic obstructive pulmonary disease. Collaborative assessment of the validity of the Tecumseh index of risk. Am Rev Respir Dis. 1984 Sep;130(3):380-5. doi: 10.1164/arrd.1984.130.3.380. PMID 6476588
- [Background] Lebowitz MD. Influence of passive smoking on pulmonary function: a survey. Prev Med. 1984 Nov;13(6):645-55. doi: 10.1016/s0091-7435(84)80014-6. PMID 6399375
- [Background] Mazzeo J, Seeley GW. A general framework for evaluating the reliability of medical measurement systems. Eval Health Prof. 1984 Dec;7(4):379-411. doi: 10.1177/016327878400700401. PMID 10269327
- [Background] Barbee RA, Dodge R, Lebowitz ML, Burrows B. The epidemiology of asthma. Chest. 1985 Jan;87(1 Suppl):21S-25S. doi: 10.1378/chest.87.1.21s. PMID 3871083
- [Background] Dodge RR, Lebowitz MD, Barbee RA, Burrows B: Immediate Reactions to Coccidioidin and Spherulin: The Relation of Atopy to Coccidioidomycosis. In: Einstein H (Ed), Coccidioidomycosis: Proceedings of the Fourth International Conference, Washington, DC: Nat'l Foundation Infectious Diseases, 1985
- [Background] Martinez F, Lebowitz MD, Taussig LM: A Longitudinal Study on the Outcome of Asthmatic Syndromes in Infancy and Childhood. Am Rev Respir Dis, 131(#4, part 2):A243, 1985
- [Background] Holberg CJ, O'Rourke MK, Lebowitz MD: A Factor For All Seasons. Am Rev Respir Dis, 131 (#4, part 2):A176, 1985
- [Background] Lebowitz MD, Holberg CJ, Boyer B, Hayes C. Respiratory symptoms and peak flow associated with indoor and outdoor air pollutants in the southwest. J Air Pollut Control Assoc. 1985 Nov;35(11):1154-8. doi: 10.1080/00022470.1985.10466016. No abstract available. PMID 4067091
- [Background] Paoletti P, Camilli AE, Holberg CJ, Lebowitz MD. Respiratory effects in relation to estimated tar exposure from current and cumulative cigarette consumption. Chest. 1985 Dec;88(6):849-55. doi: 10.1378/chest.88.6.849. PMID 4064773
- [Background] Lebowitz MD, Burrows B, Traver GA, McDonagh DJ, Dodge RR, Barbee RA, Glover J, Kennedy T, Clark D, Resar R. Methodological considerations of epidemiological diagnoses in respiratory diseases. Eur J Epidemiol. 1985 Sep;1(3):188-92. doi: 10.1007/BF00234093. PMID 3842117
- [Background] Hicks MJ, Hagaman RM, Barbee RA. The prevalence of cellular immunity to coccidioidomycosis in a highly endemic area. West J Med. 1986 Apr;144(4):425-8. PMID 3716400
- [Background] Lebowitz MD, Phibbs B, Robertson G, Holberg C, Knudson RJ, Burrows B. Vectorcardiographic and blood pressure correlates of obstructive pulmonary diseases in a community population. Chest. 1986 Jan;89(1):78-84. doi: 10.1378/chest.89.1.78. PMID 2934231
- [Background] Burrows B, Lebowitz MD, Camilli AE, Knudson RJ. Longitudinal changes in forced expiratory volume in one second in adults. Methodologic considerations and findings in healthy nonsmokers. Am Rev Respir Dis. 1986 Jun;133(6):974-80. doi: 10.1164/arrd.1986.133.6.974. PMID 3717769
- [Background] Paoletti P, Pistelli G, Fazzi P, Viegi G, Di Pede F, Giuliano G, Prediletto R, Carrozzi L, Polato R, Saetta M, et al. Reference values for vital capacity and flow-volume curves from a general population study. Bull Eur Physiopathol Respir. 1986 Sep-Oct;22(5):451-9. PMID 3492231
- [Background] Lebowitz MD: Prevalence and Natural History of Asthma. In 'Lessons From the Past' (Reed C, Ed) Bernstein IL (Ed) Guidelines for Evaluation of Nonbronchodilator Therapy of Asthma. Wash., DC: American Academy of Allergy and Immunology, pp. 8-22, 1986
- [Background] Bloom JW, Halonen M, Dunn AM, Pinnas JL, Burrows B. Pneumococcus-specific immunoglobulin E in cigarette smokers. Clin Allergy. 1986 Jan;16(1):25-32. doi: 10.1111/j.1365-2222.1986.tb01950.x. PMID 3955798
- [Background] Dodge R, Cline MG, Burrows B. Comparisons of asthma, emphysema, and chronic bronchitis diagnoses in a general population sample. Am Rev Respir Dis. 1986 Jun;133(6):981-6. doi: 10.1164/arrd.1986.133.6.981. PMID 3717770
- [Background] Bronnimann S, Burrows B. A prospective study of the natural history of asthma. Remission and relapse rates. Chest. 1986 Oct;90(4):480-4. doi: 10.1378/chest.90.4.480. PMID 3757559
- [Background] Seeley GW, Mazzeo J, Borgstrom M, Hunter TB, Newell JD, Bjelland JC. Radiologic total lung capacity measurement. Development and evaluation of a computer-based system. Eur J Radiol. 1986 Nov;6(4):262-5. PMID 3792320
- [Background] Vollmer WM, Buist AS, Johnson LR, McCamant LE, Halonen M. Relationship between serum IgE and cross-sectional and longitudinal FEV1 in two cohort studies. Chest. 1986 Sep;90(3):416-23. doi: 10.1378/chest.90.3.416. PMID 3488877
- [Background] Kibler R, Hicks MJ, Wright AL, Taussig LM. A comparative analysis of cord blood and adult lymphocytes: interleukin-2 and interferon production, natural killer cell activity, and lymphocyte populations. Diagn Immunol. 1986;4(4):201-8. PMID 2428555
- [Background] Lebowitz MD: Passive Smoking and Health Effects. In IAQ, Stockholm: Liber Tryk, 6:29-32, 1986
- [Background] Barbee RA, Kaltenborn W, Lebowitz MD, Burrows B. Longitudinal changes in allergen skin test reactivity in a community population sample. J Allergy Clin Immunol. 1987 Jan;79(1):16-24. doi: 10.1016/s0091-6749(87)80010-6. PMID 3492524
- [Background] Camilli AE, Burrows B, Knudson RJ, Lyle SK, Lebowitz MD. Longitudinal changes in forced expiratory volume in one second in adults. Effects of smoking and smoking cessation. Am Rev Respir Dis. 1987 Apr;135(4):794-9. doi: 10.1164/arrd.1987.135.4.794. PMID 3565927
- [Background] Burrows B, Knudson RJ, Camilli AE, Lyle SK, Lebowitz MD. The "horse-racing effect" and predicting decline in forced expiratory volume in one second from screening spirometry. Am Rev Respir Dis. 1987 Apr;135(4):788-93. doi: 10.1164/arrd.1987.135.4.788. PMID 3565926
- [Background] Lebowitz MD, Holberg CJ. Physiological changes in pulmonary development related to passive smoking and its interaction with active smoking. Toxicol Lett. 1987 Jan;35(1):101-5. doi: 10.1016/0378-4274(87)90092-0. PMID 3810669
- [Background] Barbee RA, Halonen M, Kaltenborn W, Lebowitz M, Burrows B. A longitudinal study of serum IgE in a community cohort: correlations with age, sex, smoking, and atopic status. J Allergy Clin Immunol. 1987 Jun;79(6):919-27. doi: 10.1016/0091-6749(87)90241-7. PMID 3584747
- [Background] Klink M, Quan SF. Prevalence of reported sleep disturbances in a general adult population and their relationship to obstructive airways diseases. Chest. 1987 Apr;91(4):540-6. doi: 10.1378/chest.91.4.540. PMID 3829746
- [Background] Knudson RJ, Kaltenborn WT, Knudson DE, Burrows B. The single-breath carbon monoxide diffusing capacity. Reference equations derived from a healthy nonsmoking population and effects of hematocrit. Am Rev Respir Dis. 1987 Apr;135(4):805-11. doi: 10.1164/arrd.1987.135.4.805. PMID 3565929
- [Background] Lebowitz MD, Holberg CJ, Knudson RJ, Burrows B. Longitudinal study of pulmonary function development in childhood, adolescence, and early adulthood. Development of pulmonary function. Am Rev Respir Dis. 1987 Jul;136(1):69-75. doi: 10.1164/ajrccm/136.1.69. PMID 3605844
- [Background] Habib MP, Klink ME, Knudson DE, Bloom JW, Kaltenborn WT, Knudson RJ. Physiologic characteristics of subjects exhibiting accelerated deterioration of ventilatory function. Am Rev Respir Dis. 1987 Sep;136(3):638-45. doi: 10.1164/ajrccm/136.3.638. PMID 3631737
- [Background] Barbee RA: The Epidemiology of Asthma. Chapter in Monograph on Epidemiology of Allergic Diseases, Schlumberger HD (Ed). S Karger, Basel, Publisher. 1987
- [Background] Lebowitz MD, Collins L, Holberg CJ. Time series analyses of respiratory responses to indoor and outdoor environmental phenomena. Environ Res. 1987 Aug;43(2):332-41. doi: 10.1016/s0013-9351(87)80033-6. PMID 3608936
- [Background] Burrows B, Bloom JW, Traver GA, Cline MG. The course and prognosis of different forms of chronic airways obstruction in a sample from the general population. N Engl J Med. 1987 Nov 19;317(21):1309-14. doi: 10.1056/NEJM198711193172103. PMID 3683459
- [Background] Holberg CJ, O'Rourke MK, Lebowitz MD. Multivariate analysis of ambient environmental factors and respiratory effects. Int J Epidemiol. 1987 Sep;16(3):399-410. doi: 10.1093/ije/16.3.399. PMID 3667038
- [Background] Lebowitz MD, Quackenboss J, Camilli AE, Bronnimann D, Holberg CJ, Boyer B. The epidemiological importance of intraindividual changes in objective pulmonary responses. Eur J Epidemiol. 1987 Dec;3(4):390-8. doi: 10.1007/BF00145651. PMID 3319671
- [Background] Quackenboss JJ, Lebowitz MD, Camilli AE, et al: Multipollutant Interactions and Health. In ibid
- [Background] Lebowitz MD, Quackenboss JJ, et al: Development of Questionnaires and Survey Instruments. In: Design and Protocol. Phila.: ASTM, (in press), 1987
- [Background] Bloom JW, Kaltenborn WT, Quan SF. Risk factors in a general population for snoring. Importance of cigarette smoking and obesity. Chest. 1988 Apr;93(4):678-83. doi: 10.1378/chest.93.4.678. PMID 3258226
- [Background] Burrows B, Knudson RJ, Cline MG, Lebowitz MD. A reexamination of risk factors for ventilatory impairment. Am Rev Respir Dis. 1988 Oct;138(4):829-36. doi: 10.1164/ajrccm/138.4.829. PMID 3202457
- [Background] Lebowitz MD: Respiratory Symptom: Concepts and Techniques for the Study of Respiratory Changes in Aging. In: Kent B and Butler RN (Eds), Human Aging Research: Concepts and Techniques. New York: Raven Press, 1988
- [Background] Lebowitz MD, Holberg CJ. Effects of parental smoking and other risk factors on the development of pulmonary function in children and adolescents. Analysis of two longitudinal population studies. Am J Epidemiol. 1988 Sep;128(3):589-97. doi: 10.1093/oxfordjournals.aje.a115006. PMID 3414663
- [Background] Lebowitz MD: Prevalence and Incidence Rates of Airway Obstructive Peroblems: An International Comparison. Med Thoracica, 10:189-93, 1988
- [Background] Lebowitz MD: Allergy Sufferers in the Southwest. Medical and Health Annual Chicago: Encyclopedia Britannica, pp. 274-276, 1988
- [Background] Burrows B, Martinez FD, Halonen M, Barbee RA, Cline MG. Association of asthma with serum IgE levels and skin-test reactivity to allergens. N Engl J Med. 1989 Feb 2;320(5):271-7. doi: 10.1056/NEJM198902023200502. PMID 2911321
- [Background] Burrows B: Distribution of Allergy in the General Population. In: Bronchits IV. Proceedings Royal Van Gorcum Assen. The Netherlands. pp. 3-13, 1989
- [Background] Burrows B: Allergy and Its Relationship to Asthma, Bronchial Reactivity and Chronic Airways Obstruction: An Epidemiological Perspective. In: S.T. Weiss and D. Sparrow (Eds), Airways Responsiveness and Allergy in the Development of Chronic Lung Disease. Raven Press, New York, NY, pp. 241-270, 1989
- [Background] Barbee RA: Airways Responsiveness and Allergy in the Development of Chronic Lung Disease. In: Methodological Issues in the Assessment of Allergy. Edited by ST Weiss, M.D. and D Sparrow, M.D. Raven Press, New York, 1989
- [Background] Burrows B: Natural History of Chronic Airflow Obstruction. In: Clinical Epidemiology of Chronic Obstructive Pulmonary Disease (Eds) M Hensley and NA Saunders. Marcel Dekker, Inc., 1989
- [Background] Sherrill DL, Morgan WJ, Taussig LM, Landau LI, Burrows B. A mathematical procedure for estimating the spatial relationships between lung function, somatic growth, and maturation. Pediatr Res. 1989 Mar;25(3):316-21. doi: 10.1203/00006450-198903000-00022. PMID 2704599
- [Background] Cline MG, Burrows B. Distribution of allergy in a population sample residing in Tucson, Arizona. Thorax. 1989 May;44(5):425-31. doi: 10.1136/thx.44.5.425. No abstract available. PMID 2763244
- [Background] Cline MG, Meredith KE, Boyer JT, Burrows B. Decline of height with age in adults in a general population sample: estimating maximum height and distinguishing birth cohort effects from actual loss of stature with aging. Hum Biol. 1989 Jun;61(3):415-25. PMID 2807265
- [Background] Lebowitz MD. The trends in airway obstructive disease morbidity in the Tucson Epidemiological Study. Am Rev Respir Dis. 1989 Sep;140(3 Pt 2):S35-41. doi: 10.1164/ajrccm/140.3_Pt_2.S35. PMID 2782758
- [Background] Sherrill DL, Camilli A, Lebowitz MD. On the temporal relationships between lung function and somatic growth. Am Rev Respir Dis. 1989 Sep;140(3):638-44. doi: 10.1164/ajrccm/140.3.638. PMID 2782737
- [Background] McGue M, Gerrard JW, Lebowitz MD, Rao DC. Commingling in the distributions of immunoglobulin levels. Hum Hered. 1989;39(4):196-201. doi: 10.1159/000153860. PMID 2583731
- [Background] Knudson RJ, Kaltenborn WT, Burrows B. The effects of cigarette smoking and smoking cessation on the carbon monoxide diffusing capacity of the lung in asymptomatic subjects. Am Rev Respir Dis. 1989 Sep;140(3):645-51. doi: 10.1164/ajrccm/140.3.645. PMID 2782738
- [Background] Burrows B. The course and prognosis of different types of chronic airflow limitation in a general population sample from Arizona: comparison with the Chicago "COPD" series. Am Rev Respir Dis. 1989 Sep;140(3 Pt 2):S92-4. doi: 10.1164/ajrccm/140.3_Pt_2.S92. PMID 2782767
- [Background] Paoletti P, Prediletto R, Carrozzi L, Viegi G, Di Pede F, Carmignani G, Mammini U, Giuntini C, Lebowitz MD. Effects of childhood and adolescence-adulthood respiratory infections in a general population. Eur Respir J. 1989 May;2(5):428-36. PMID 2788099
- [Background] Krzyzanowski M, Sherrill DL, Lebowitz MD. Longitudinal analysis of the effects of acute lower respiratory illnesses on pulmonary function in an adult population. Am J Epidemiol. 1990 Mar;131(3):412-22. doi: 10.1093/oxfordjournals.aje.a115516. PMID 2301351
- [Background] Sherrill D, Holberg CJ, Lebowitz MD. Differential rates of lung growth as measured longitudinally by pulmonary function in children and adolescents. Pediatr Pulmonol. 1990;8(3):145-54. doi: 10.1002/ppul.1950080304. PMID 2349006
- [Background] Krzyzanowski M, Camilli AE, Lebowitz MD. Relationships between pulmonary function and changes in chronic respiratory symptoms. Comparison of Tucson and Cracow longitudinal studies. Chest. 1990 Jul;98(1):62-70. doi: 10.1378/chest.98.1.62. PMID 2361414
- [Background] Lebowitz MD, Holberg CJ. Comparisons of spirometric reference values and the proportions of abnormal subjects among male smokers and those symptomatic in a community population. Am Rev Respir Dis. 1990 Jun;141(6):1491-6. doi: 10.1164/ajrccm/141.6.1491. PMID 2350090
- [Background] Burrows B. Airways obstructive diseases: pathogenetic mechanisms and natural histories of the disorders. Med Clin North Am. 1990 May;74(3):547-59. doi: 10.1016/s0025-7125(16)30539-9. PMID 2186232
- [Background] Viegi G, Paoletti P, Prediletto R, Di Pede F, Carrozzi L, Carmignani G, Mammini U, Lebowitz MD, Giuntini C. Carbon monoxide diffusing capacity, other indices of lung function, and respiratory symptoms in a general population sample. Am Rev Respir Dis. 1990 Apr;141(4 Pt 1):1033-9. doi: 10.1164/ajrccm/141.4_Pt_1.1033. PMID 2327637
- [Background] Barbee RA, Halonen M, Kaltenborn WT, Burrows B. A longitudinal study of respiratory symptoms in a community population sample. Correlations with smoking, allergen skin-test reactivity, and serum IgE. Chest. 1991 Jan;99(1):20-6. doi: 10.1378/chest.99.1.20. PMID 1984955
- [Background] John TJ, Sieber OF Jr. Chemotactic migration of neutrophils under agarose. Life Sci. 1976 Jan 15;18(2):177-81. doi: 10.1016/0024-3205(76)90022-9. No abstract available. PMID 1256233
- [Background] Sieber OF Jr, Lucas DL, Lohman C, Larter W, Giles H, John TJ: Reactivity of Lymphocytes in Maternal and Cord Blood to Respiratory Syncytial Virus. Clin Res, XXIV, 181A, 1976
- [Background] Strunk RC, Sieber OF, Taussig LM, Gall EP. Serum complement depression during viral lower respiratory tract illness in cystic fibrosis. Arch Dis Child. 1977 Sep;52(9):687-90. doi: 10.1136/adc.52.9.687. PMID 921318
- [Background] Taussig LM, Harris TR, Lebowitz MD. Lung function in infants and young children: functional residual capacity, tidal volume, and respiratory rats. Am Rev Respir Dis. 1977 Aug;116(2):233-9. doi: 10.1164/arrd.1977.116.2.233. PMID 889175
- [Background] Taussig LM. Maximal expiratory flows at functional residual capacity: a test of lung function for young children. Am Rev Respir Dis. 1977 Dec;116(6):1031-8. doi: 10.1164/arrd.1977.116.6.1031. PMID 931179
- [Background] Ellis EF. Relationship between the allergic state and susceptibility to infectious airway disease. Pediatr Res. 1977 Mar;11(3 Pt 2):227-9. No abstract available. PMID 322073
- [Background] Taussig LM. Clinical and physiologic evidence for the persistence of pulmonary abnormalities after respiratory illnesses in infancy and childhood. Pediatr Res. 1977 Mar;11(3 Pt 2):216-8. No abstract available. PMID 322072
- [Background] Feldman J, Traver GA, Taussig LM. Maximal expiratory flows after postural drainage. Am Rev Respir Dis. 1979 Feb;119(2):239-45. doi: 10.1164/arrd.1979.119.2.239. PMID 434596
- [Background] Harrison HR, Riggin RT. Infection of untreated primary human amnion monolayers with Chlamydia trachomatis. J Infect Dis. 1979 Dec;140(6):968-71. doi: 10.1093/infdis/140.6.968. PMID 541524
- [Background] Nickerson BG, Taussig LM. Family history of asthma in infants with bronchopulmonary dysplasia. Pediatrics. 1980 Jun;65(6):1140-4. PMID 7375238
- [Background] Loughlin GM, Cota KA, Taussig LM. The relationship between flow transients and bronchial lability in cystic fibrosis. Chest. 1981 Feb;79(2):206-10. doi: 10.1378/chest.79.2.206. PMID 7460652
- [Background] Nickerson BG, Lemen RJ, Gerdes CB, Wegmann MJ, Robertson G. Within-subject variability and per cent change for significance of spirometry in normal subjects and in patients with cystic fibrosis. Am Rev Respir Dis. 1980 Dec;122(6):859-66. doi: 10.1164/arrd.1980.122.6.859. PMID 7458059
- [Background] Wagener JS, Taussig LM, DeBenedetti C, Lemen RJ, Loughlin GM. Pulmonary function in juvenile rheumatoid arthritis. J Pediatr. 1981 Jul;99(1):108-10. doi: 10.1016/s0022-3476(81)80972-9. No abstract available. PMID 7252647
- [Background] Taussig LM, Smith SM, Blumenfeld R. Chronic bronchitis in childhood: what is it? Pediatrics. 1981 Jan;67(1):1-5. PMID 7243418
- [Background] Taussig LM, Cota K, Kaltenborn W. Different mechanical properties of the lung in boys and girls. Am Rev Respir Dis. 1981 Jun;123(6):640-3. doi: 10.1164/arrd.1981.123.6.640. PMID 7271061
- [Background] Manthei U, Taussig LM, Beckerman RC, Strunk RC. Circulating immune complexes in cystic fibrosis. Am Rev Respir Dis. 1982 Aug;126(2):253-7. doi: 10.1164/arrd.1982.126.2.253. PMID 7103251
- [Background] Taussig LM, Landau LI, Godfrey S, Arad I. Determinants of forced expiratory flows in newborn infants. J Appl Physiol Respir Environ Exerc Physiol. 1982 Nov;53(5):1220-7. doi: 10.1152/jappl.1982.53.5.1220. PMID 7174416
- [Background] Harrison HR, Taussig LM, Fulginiti VA. Chlamydia trachomatis and chronic respiratory disease in childhood. Pediatr Infect Dis. 1982 Jan-Feb;1(1):29-33. doi: 10.1097/00006454-198201000-00008. PMID 7177892
- [Background] Sobonya RE, Logvinoff MM, Taussig LM, Theriault A. Morphometric analysis of the lung in prolonged bronchopulmonary dysplasia. Pediatr Res. 1982 Nov;16(11):969-72. doi: 10.1203/00006450-198211000-00014. PMID 7155668
- [Background] Godfrey S, Bar-Yishay E, Arad I, Landau LI, Taussig LM. Flow-volume curves in infants with lung disease. Pediatrics. 1983 Oct;72(4):517-22. PMID 6889065
- [Background] Davis PB, Hubbard VS, McCoy K, Taussig LM. Familial bronchiectasis. J Pediatr. 1983 Feb;102(2):177-85. doi: 10.1016/s0022-3476(83)80515-0. No abstract available. PMID 6822919
- [Background] Logvinoff MM, Fon GT, Taussig LM, Pitt MJ. Kyphosis and pulmonary function in cystic fibrosis. Clin Pediatr (Phila). 1984 Jul;23(7):389-92. doi: 10.1177/000992288402300705. PMID 6723186
- [Background] Pagtakhan RD, Bjelland JC, Landau LI, Loughlin G, Kaltenborn W, Seeley G, Taussig LM. Sex differences in growth patterns of the airways and lung parenchyma in children. J Appl Physiol Respir Environ Exerc Physiol. 1984 May;56(5):1204-10. doi: 10.1152/jappl.1984.56.5.1204. PMID 6725083
- [Background] Tepper RS, Pagtakhan RD, Taussig LM. Noninvasive determination of total respiratory system compliance in infants by the weighted-spirometer method. Am Rev Respir Dis. 1984 Sep;130(3):461-6. doi: 10.1164/arrd.1984.130.3.461. PMID 6383155
- [Background] Morgan WJ, Taussig LM. The chronic bronchitis complex in children. Pediatr Clin North Am. 1984 Aug;31(4):851-64. doi: 10.1016/s0031-3955(16)34649-1. PMID 6146959
- [Background] Soto ME, Sly PD, Uren E, Taussig LM, Landau LI. Bronchodilator response during acute viral bronchiolitis in infancy. Pediatr Pulmonol. 1985 Mar-Apr;1(2):85-90. doi: 10.1002/ppul.1950010206. PMID 4069797
- [Background] Reiter EO, Brugman SM, Pike JW, Pitt M, Dokoh S, Haussler MR, Gerstle RS, Taussig LM. Vitamin D metabolites in adolescents and young adults with cystic fibrosis: effects of sun and season. J Pediatr. 1985 Jan;106(1):21-6. doi: 10.1016/s0022-3476(85)80458-3. PMID 3871230
- [Background] Carroll J, Taussig LM: Pulmonary Disorders. In: Immunologic Disorders in Infants and Children. Stiehm ER (Ed). W. B. Saunders Co. Edition III, 1985
- [Background] Sobonya RE, Taussig LM. Quantitative aspects of lung pathology in cystic fibrosis. Am Rev Respir Dis. 1986 Aug;134(2):290-5. doi: 10.1164/arrd.1986.134.2.290. PMID 3740655
- [Background] Tepper RS, Morgan WJ, Cota K, Wright A, Taussig LM. Physiologic growth and development of the lung during the first year of life. Am Rev Respir Dis. 1986 Sep;134(3):513-9. doi: 10.1164/arrd.1986.134.3.513. PMID 3752707
- [Background] Tepper RS, Morgan WJ, Cota K, Taussig LM. Expiratory flow limitation in infants with bronchopulmonary dysplasia. J Pediatr. 1986 Dec;109(6):1040-6. doi: 10.1016/s0022-3476(86)80296-7. PMID 3783328
- [Background] Schumacher MJ, Cota KA, Taussig LM. Pulmonary response to nasal-challenge testing of atopic subjects with stable asthma. J Allergy Clin Immunol. 1986 Jul;78(1 Pt 1):30-5. doi: 10.1016/0091-6749(86)90111-9. PMID 3722633
- [Background] Mellins R, Chernick V, Clyde W, Farrell P, Glezen WP, Rigatto H, Taussig LM: Pediatric Respiratory Disorders. NIH Publication #86-2107 August 1986
- [Background] Morgan WJ, Taussig LM. The child with persistent cough. Pediatr Rev. 1987 Feb;8(8):249-53. doi: 10.1542/pir.8-8-249. No abstract available. PMID 3332355
- [Background] Smith JJ, Lemen RJ, Taussig LM. Mechanisms of viral-induced lower airway obstruction. Pediatr Infect Dis J. 1987 Sep;6(9):837-42. doi: 10.1097/00006454-198709000-00010. No abstract available. PMID 3313249
- [Background] Martinez FD, Morgan WJ, Wright AL, Holberg CJ, Taussig LM. Diminished lung function as a predisposing factor for wheezing respiratory illness in infants. N Engl J Med. 1988 Oct 27;319(17):1112-7. doi: 10.1056/NEJM198810273191702. PMID 3173442
- [Background] Morgan WJ, Geller DE, Tepper RS, Taussig LM. Partial expiratory flow-volume curves in infants and young children. Pediatr Pulmonol. 1988;5(4):232-43. doi: 10.1002/ppul.1950050410. No abstract available. PMID 3070472
- [Background] Wright AL, Holberg C, Taussig LM. Infant-feeding practices among middle-class Anglos and Hispanics. Pediatrics. 1988 Sep;82(3 Pt 2):496-503. PMID 3405686
- [Background] Geller DE, Morgan WJ, Cota KA, Wright AL, Taussig LM. Airway responsiveness to cold, dry air in normal infants. Pediatr Pulmonol. 1988;4(2):90-7. doi: 10.1002/ppul.1950040206. PMID 3380581
- [Background] Morgan WJ: Evaluation of Forced Expiratory Flow in Infants. Proceedings of the Second State of the Art Conference on Neonatal Pulmonary Function Testing, Chicago, Perinatology Press, Ithaca, NY, 1988
- [Background] Wright AL. Models of mystery: physician and patient perceptions of sudden infant death syndrome. Soc Sci Med. 1988;26(6):587-95. doi: 10.1016/0277-9536(88)90022-6. PMID 3363400
- [Background] Humphries CT, Wagener JS, Morgan WJ. Fatal prolonged foreign body aspiration following an asymptomatic interval. Am J Emerg Med. 1988 Nov;6(6):611-3. doi: 10.1016/0735-6757(88)90104-0. PMID 3178959
- [Background] Taussig LM, Wright AL, Morgan WJ, Harrison HR, Ray CG. The Tucson Children's Respiratory Study. I. Design and implementation of a prospective study of acute and chronic respiratory illness in children. Am J Epidemiol. 1989 Jun;129(6):1219-31. doi: 10.1093/oxfordjournals.aje.a115242. PMID 2729258
- [Background] Wright AL, Taussig LM, Ray CG, Harrison HR, Holberg CJ. The Tucson Children's Respiratory Study. II. Lower respiratory tract illness in the first year of life. Am J Epidemiol. 1989 Jun;129(6):1232-46. doi: 10.1093/oxfordjournals.aje.a115243. PMID 2729259
- [Background] Wright AL, Holberg CJ, Martinez FD, Morgan WJ, Taussig LM. Breast feeding and lower respiratory tract illness in the first year of life. Group Health Medical Associates. BMJ. 1989 Oct 14;299(6705):946-9. doi: 10.1136/bmj.299.6705.946. PMID 2508946
- [Background] Boyce WT, Schaefer C, Harrison HR, Haffner WH, Lewis M, Wright AL. Sociocultural factors in puerperal infectious morbidity among Navajo women. Am J Epidemiol. 1989 Mar;129(3):604-15. doi: 10.1093/oxfordjournals.aje.a115173. PMID 2916554
- [Background] Hoit JD, Hixon TJ, Altman ME, Morgan WJ. Speech breathing in women. J Speech Hear Res. 1989 Jun;32(2):353-65. doi: 10.1044/jshr.3202.353. PMID 2739388
- [Background] Neddenriep D, Taussig LM: Infection of the Lower Respiratory Tract. In: Enchenwald, HF (Ed), Current Therapy in Pediatrics, 2, B.C. Decker Co, 1989
- [Background] Summut PH, Taussig LM: Cystic Fibrosis in the Adolescent and Adult. In: Current Pulmonolgy, Vol. 10, Year Book Medical Publishers, 1989
- [Background] Grad R, Taussig LM: Acute Infections Producing Upper Airway Obstruction. In: Chernick, V (Ed): Disorders of the Respiratory Tract in Children, 5th Ed., Saunders Co., 1989
- [Background] Martinez FD, Taussig LM, Morgan WJ. Infants with upper respiratory illnesses have significant reductions in maximal expiratory flow. Pediatr Pulmonol. 1990;9(2):91-5. doi: 10.1002/ppul.1950090206. PMID 2399052
- [Background] Wright AL, Morgan WJ. On the creation of 'problem' patients. Soc Sci Med. 1990;30(9):951-9. doi: 10.1016/0277-9536(90)90142-f. PMID 2336573
- [Background] Martinez FD, Wright AL, Holberg CJ, Morgan WJ, Taussig LM. Maternal age as a risk factor for wheezing lower respiratory illnesses in the first year of life. Am J Epidemiol. 1992 Nov 15;136(10):1258-68. doi: 10.1093/oxfordjournals.aje.a116434. PMID 1476148
- [Background] Morgan WJ, Martinez FD. Risk factors for developing wheezing and asthma in childhood. Pediatr Clin North Am. 1992 Dec;39(6):1185-203. doi: 10.1016/s0031-3955(16)38440-1. PMID 1437315
- [Background] Halonen M, Stern D, Taussig LM, Wright A, Ray CG, Martinez FD. The predictive relationship between serum IgE levels at birth and subsequent incidences of lower respiratory illnesses and eczema in infants. Am Rev Respir Dis. 1992 Oct;146(4):866-70. doi: 10.1164/ajrccm/146.4.866. PMID 1416412
- [Background] Burrows B, Sears MR, Flannery EM, Herbison GP, Holdaway MD. Relationships of bronchial responsiveness assessed by methacholine to serum IgE, lung function, symptoms, and diagnoses in 11-year-old New Zealand children. J Allergy Clin Immunol. 1992 Sep;90(3 Pt 1):376-85. doi: 10.1016/s0091-6749(05)80018-1. PMID 1527320
- [Background] Klink ME, Quan SF, Kaltenborn WT, Lebowitz MD. Risk factors associated with complaints of insomnia in a general adult population. Influence of previous complaints of insomnia. Arch Intern Med. 1992 Aug;152(8):1634-7. PMID 1497397
- [Background] Sherrill D, Sears MR, Lebowitz MD, Holdaway MD, Hewitt CJ, Flannery EM, Herbison GP, Silva PA. The effects of airway hyperresponsiveness, wheezing, and atopy on longitudinal pulmonary function in children: a 6-year follow-up study. Pediatr Pulmonol. 1992 Jun;13(2):78-85. doi: 10.1002/ppul.1950130204. PMID 1495861
- [Background] Stern DA, Hicks MJ, Martinez FD, Holberg CJ, Wright AL, Pinnas J, Halonen M, Taussig LM. Lymphocyte subpopulation number and function in infancy. Dev Immunol. 1992;2(3):175-9. doi: 10.1155/1992/64292. PMID 1627949
- [Background] Lebowitz MD, Sherrill D, Holberg CJ. Effects of passive smoking on lung growth in children. Pediatr Pulmonol. 1992 Jan;12(1):37-42. doi: 10.1002/ppul.1950120109. PMID 1579375
- [Background] Krzyzanowski M, Lebowitz MD. Changes in chronic respiratory symptoms in two populations of adults studied longitudinally over 13 years. Eur Respir J. 1992 Jan;5(1):12-20. PMID 1577133
- [Background] Witten ML, Grad R, Quan SF, Lantz RC, Sobonya RE, Lemen RJ. Effects of respiratory viruses on pulmonary alveolar macrophages. Pediatr Pulmonol. 1992 Feb;12(2):105-12. doi: 10.1002/ppul.1950120209. No abstract available. PMID 1570188
- [Background] Sherrill DL, Lebowitz MD, Knudson RJ, Burrows B. Continuous longitudinal regression equations for pulmonary function measures. Eur Respir J. 1992 Apr;5(4):452-62. PMID 1563504
- [Background] Martinez FD, Cline M, Burrows B. Increased incidence of asthma in children of smoking mothers. Pediatrics. 1992 Jan;89(1):21-6. PMID 1728015
- [Background] Lebowitz MD. The use of peak expiratory flow rate measurements in respiratory disease. Pediatr Pulmonol. 1991;11(2):166-74. doi: 10.1002/ppul.1950110215. No abstract available. PMID 1758735
- [Background] Burrows B, Lebowitz MD, Barbee RA, Cline MG. Findings before diagnoses of asthma among the elderly in a longitudinal study of a general population sample. J Allergy Clin Immunol. 1991 Dec;88(6):870-7. doi: 10.1016/0091-6749(91)90243-h. PMID 1744357
- [Background] Burrows B, Barbee RA, Cline MG, Knudson RJ, Lebowitz MD. Characteristics of asthma among elderly adults in a sample of the general population. Chest. 1991 Oct;100(4):935-42. doi: 10.1378/chest.100.4.935. PMID 1914608
- [Background] Sears MR, Burrows B, Flannery EM, Herbison GP, Hewitt CJ, Holdaway MD. Relation between airway responsiveness and serum IgE in children with asthma and in apparently normal children. N Engl J Med. 1991 Oct 10;325(15):1067-71. doi: 10.1056/NEJM199110103251504. PMID 1891008
- [Background] Sherrill DL, Krzyzanowski M, Bloom JW, Lebowitz MD. Respiratory effects of non-tobacco cigarettes: a longitudinal study in general population. Int J Epidemiol. 1991 Mar;20(1):132-7. doi: 10.1093/ije/20.1.132. PMID 2066211
- [Background] Sherrill DL, Lebowitz MD, Knudson RJ, Burrows B. Smoking and symptom effects on the curves of lung function growth and decline. Am Rev Respir Dis. 1991 Jul;144(1):17-22. doi: 10.1164/ajrccm/144.1.17. PMID 2064125
- [Background] Burrows B. Epidemiologic evidence for different types of chronic airflow obstruction. Am Rev Respir Dis. 1991 Jun;143(6):1452-4; discussion 1455. doi: 10.1164/ajrccm/143.6.1452. No abstract available. PMID 2048836
- [Background] Halonen M, Stern D, Lyle S, Wright A, Taussig L, Martinez FD. Relationship of total serum IgE levels in cord and 9-month sera of infants. Clin Exp Allergy. 1991 Mar;21(2):235-41. doi: 10.1111/j.1365-2222.1991.tb00836.x. PMID 2043992
- [Background] Knudson RJ, Standen JR, Kaltenborn WT, Knudson DE, Rehm K, Habib MP, Newell JD. Expiratory computed tomography for assessment of suspected pulmonary emphysema. Chest. 1991 Jun;99(6):1357-66. doi: 10.1378/chest.99.6.1357. PMID 2036816
- [Background] Holberg CJ, Wright AL, Martinez FD, Ray CG, Taussig LM, Lebowitz MD. Risk factors for respiratory syncytial virus-associated lower respiratory illnesses in the first year of life. Am J Epidemiol. 1991 Jun 1;133(11):1135-51. doi: 10.1093/oxfordjournals.aje.a115826. PMID 2035517
- [Background] Camilli AE, Robbins DR, Lebowitz MD. Death certificate reporting of confirmed airways obstructive disease. Am J Epidemiol. 1991 Apr 15;133(8):795-800. doi: 10.1093/oxfordjournals.aje.a115958. PMID 2021146
- [Background] Quackenboss JJ, Lebowitz MD, Krzyzanowski M. The normal range of diurnal changes in peak expiratory flow rates. Relationship to symptoms and respiratory disease. Am Rev Respir Dis. 1991 Feb;143(2):323-30. doi: 10.1164/ajrccm/143.2.323. PMID 1990947
- [Background] Krzyzanowski M, Sherrill DL, Paoletti P, Lebowitz MD. Relationship of respiratory symptoms and pulmonary function to tar, nicotine, and carbon monoxide yield of cigarettes. Am Rev Respir Dis. 1991 Feb;143(2):306-11. doi: 10.1164/ajrccm/143.2.306. PMID 1990944
- [Background] Lebowitz MD, Holberg CJ, Martinez FD. A longitudinal study of risk factors in asthma and chronic bronchitis in childhood. Eur J Epidemiol. 1990 Dec;6(4):341-7. doi: 10.1007/BF00151706. PMID 2091933
- [Background] Burrows B. Differential diagnosis of chronic obstructive pulmonary disease. Chest. 1990 Feb;97(2 Suppl):16S-18S. doi: 10.1378/chest.97.2_supplement.16s. PMID 2404707
- [Background] Klink M, Cline MG, Halonen M, Burrows B. Problems in defining normal limits for serum IgE. J Allergy Clin Immunol. 1990 Feb;85(2):440-4. doi: 10.1016/0091-6749(90)90153-u. PMID 2303647
- [Background] Martinez FD, Holberg CJ. Segregation analysis of physician-diagnosed asthma in Hispanic and non-Hispanic white families. Clin Exp Allergy. 1995 Nov;25 Suppl 2:68-70; discussion 95-6. No abstract available. PMID 8590348
- [Background] Lebowitz MD, Bronnimann S, Camilli AE. Asthmatic risk factors and bronchial reactivity in non-diagnosed asthmatic adults. Eur J Epidemiol. 1995 Oct;11(5):541-8. doi: 10.1007/BF01719306. PMID 8549728
- [Background] Martinez FD, Stern DA, Wright AL, Holberg CJ, Taussig LM, Halonen M. Association of interleukin-2 and interferon-gamma production by blood mononuclear cells in infancy with parental allergy skin tests and with subsequent development of atopy. J Allergy Clin Immunol. 1995 Nov;96(5 Pt 1):652-60. doi: 10.1016/s0091-6749(95)70264-4. PMID 7499682
- [Background] Martinez FD, Stern DA, Wright AL, Taussig LM, Halonen M. Association of non-wheezing lower respiratory tract illnesses in early life with persistently diminished serum IgE levels. Group Health Medical Associates. Thorax. 1995 Oct;50(10):1067-72. doi: 10.1136/thx.50.10.1067. PMID 7491555
- [Background] Burrows B, Martinez FD, Cline MG, Lebowitz MD. The relationship between parental and children's serum IgE and asthma. Am J Respir Crit Care Med. 1995 Nov;152(5 Pt 1):1497-500. doi: 10.1164/ajrccm.152.5.7582283.
- [Background] Burrows B, Sears MR, Flannery EM, Herbison GP, Holdaway MD, Silva PA. Relation of the course of bronchial responsiveness from age 9 to age 15 to allergy. Am J Respir Crit Care Med. 1995 Oct;152(4 Pt 1):1302-8. doi: 10.1164/ajrccm.152.4.7551386.
- [Background] Lebowitz MD, Sherrill DL. The assessment and interpretation of spirometry during the transition from childhood to adulthood. Pediatr Pulmonol. 1995 Feb;19(2):143-9. doi: 10.1002/ppul.1950190210. No abstract available. PMID 7659470
- [Background] von Mutius E, Sherrill DL, Fritzsch C, Martinez FD, Lebowitz MD. Air pollution and upper respiratory symptoms in children from East Germany. Eur Respir J. 1995 May;8(5):723-8. PMID 7656942
- [Background] Honsberg AE, Dodge RR, Cline MG, Quan SF. Incidence and remission of habitual snoring over a 5- to 6-year period. Chest. 1995 Sep;108(3):604-9. doi: 10.1378/chest.108.3.604. PMID 7656604
- [Background] Dodge R, Cline MG, Quan SF. The natural history of insomnia and its relationship to respiratory symptoms. Arch Intern Med. 1995 Sep 11;155(16):1797-800. PMID 7654114
- [Background] Lebowitz MD, Postma DS, Burrows B. Adverse effects of eosinophilia and smoking on the natural history of newly diagnosed chronic bronchitis. Chest. 1995 Jul;108(1):55-61. doi: 10.1378/chest.108.1.55. PMID 7606992
- [Background] Sherrill DL, Lebowitz MD, Halonen M, Barbee RA, Burrows B. Longitudinal evaluation of the association between pulmonary function and total serum IgE. Am J Respir Crit Care Med. 1995 Jul;152(1):98-102. doi: 10.1164/ajrccm.152.1.7599870.
- [Background] Postma DS, Lebowitz MD. Persistence and new onset of asthma and chronic bronchitis evaluated longitudinally in a community population sample of adults. Arch Intern Med. 1995 Jul 10;155(13):1393-9. PMID 7794088
- [Background] Ey JL, Holberg CJ, Aldous MB, Wright AL, Martinez FD, Taussig LM. Passive smoke exposure and otitis media in the first year of life. Group Health Medical Associates. Pediatrics. 1995 May;95(5):670-7. PMID 7724301
- [Background] Witt-Enderby PA, Yamamura HI, Halonen M, Lai J, Palmer JD, Bloom JW. Regulation of airway muscarinic cholinergic receptor subtypes by chronic anticholinergic treatment. Mol Pharmacol. 1995 Mar;47(3):485-90. PMID 7700247
- [Background] Burrows B, Sears MR, Flannery EM, Herbison GP, Holdaway MD. Relations of bronchial responsiveness to allergy skin test reactivity, lung function, respiratory symptoms, and diagnoses in thirteen-year-old New Zealand children. J Allergy Clin Immunol. 1995 Feb;95(2):548-56. doi: 10.1016/s0091-6749(95)70317-9. PMID 7852671
- [Background] Martinez FD, Wright AL, Taussig LM, Holberg CJ, Halonen M, Morgan WJ. Asthma and wheezing in the first six years of life. The Group Health Medical Associates. N Engl J Med. 1995 Jan 19;332(3):133-8. doi: 10.1056/NEJM199501193320301. PMID 7800004
- [Background] Sherrill DL, Halonen M, Burrows B. Relationships between total serum IgE, atopy, and smoking: a twenty-year follow-up analysis. J Allergy Clin Immunol. 1994 Dec;94(6 Pt 1):954-62. doi: 10.1016/0091-6749(94)90113-9. PMID 7798543
- [Background] Dodge R, Cline MG, Lebowitz MD, Burrows B. Findings before the diagnosis of asthma in young adults. J Allergy Clin Immunol. 1994 Nov;94(5):831-5. doi: 10.1016/0091-6749(94)90150-3. PMID 7963152
- [Background] Cline MG, Dodge R, Lebowitz MD, Burrows B. Determinants of percent predicted FEV1 in current asthmatic subjects. Chest. 1994 Oct;106(4):1089-93. doi: 10.1378/chest.106.4.1089. PMID 7924478
- [Background] Martinez FD, Wright AL, Taussig LM. The effect of paternal smoking on the birthweight of newborns whose mothers did not smoke. Group Health Medical Associates. Am J Public Health. 1994 Sep;84(9):1489-91. doi: 10.2105/ajph.84.9.1489. PMID 8092378
- [Background] Martinez FD, Holberg CJ, Halonen M, Morgan WJ, Wright AL, Taussig LM. Evidence for Mendelian inheritance of serum IgE levels in Hispanic and non-Hispanic white families. Am J Hum Genet. 1994 Sep;55(3):555-65. PMID 8079994
- [Background] von Mutius E, Martinez FD, Fritzsch C, Nicolai T, Reitmeir P, Thiemann HH. Skin test reactivity and number of siblings. BMJ. 1994 Mar 12;308(6930):692-5. doi: 10.1136/bmj.308.6930.692. PMID 8142793
- [Background] Sherrill DL, Holberg CJ, Enright PL, Lebowitz MD, Burrows B. Longitudinal analysis of the effects of smoking onset and cessation on pulmonary function. Am J Respir Crit Care Med. 1994 Mar;149(3 Pt 1):591-7. doi: 10.1164/ajrccm.149.3.8118623.
- [Background] von Mutius E, Martinez FD, Fritzsch C, Nicolai T, Roell G, Thiemann HH. Prevalence of asthma and atopy in two areas of West and East Germany. Am J Respir Crit Care Med. 1994 Feb;149(2 Pt 1):358-64. doi: 10.1164/ajrccm.149.2.8306030.
- [Background] Klink ME, Dodge R, Quan SF. The relation of sleep complaints to respiratory symptoms in a general population. Chest. 1994 Jan;105(1):151-4. doi: 10.1378/chest.105.1.151. PMID 8275723
- [Background] Camilli AE, Holberg CJ, Wright AL, Taussig LM. Parental childhood respiratory illness and respiratory illness in their infants. Group Health Medical Associates. Pediatr Pulmonol. 1993 Nov;16(5):275-80. doi: 10.1002/ppul.1950160502. PMID 8255631
- [Background] Dodge R, Burrows B, Lebowitz MD, Cline MG. Antecedent features of children in whom asthma develops during the second decade of life. J Allergy Clin Immunol. 1993 Nov;92(5):744-9. doi: 10.1016/0091-6749(93)90018-b. PMID 8227866
- [Background] von Mutius E, Nicolai T, Martinez FD. Prematurity as a risk factor for asthma in preadolescent children. J Pediatr. 1993 Aug;123(2):223-9. doi: 10.1016/s0022-3476(05)81692-0. PMID 8345417
- [Background] Holberg CJ, Wright AL, Martinez FD, Morgan WJ, Taussig LM. Child day care, smoking by caregivers, and lower respiratory tract illness in the first 3 years of life. Group Health Medical Associates. Pediatrics. 1993 May;91(5):885-92. PMID 8474807
- [Background] Krzyzanowski M, Robbins DR, Lebowitz MD. Smoking cessation and changes in respiratory symptoms in two populations followed for 13 years. Int J Epidemiol. 1993 Aug;22(4):666-73. doi: 10.1093/ije/22.4.666. PMID 8225741
- [Background] Sherrill DL, Martinez FD, Sears MR, Lebowitz MD. An alternative method for comparing and describing methacholine response curves. Am Rev Respir Dis. 1993 Jul;148(1):116-22. doi: 10.1164/ajrccm/148.1.116. PMID 8317786
- [Background] Wright AL, Holberg CJ, Taussig LM, Martinez FD. Relationship of infant feeding to recurrent wheezing at age 6 years. Arch Pediatr Adolesc Med. 1995 Jul;149(7):758-63. doi: 10.1001/archpedi.1995.02170200048006. PMID 7795765
- [Background] Wright AL, Holberg CJ, Martinez FD, Halonen M, Morgan W, Taussig LM. Epidemiology of physician-diagnosed allergic rhinitis in childhood. Pediatrics. 1994 Dec;94(6 Pt 1):895-901. PMID 7971008
- [Background] Ray CG, Holberg CJ, Minnich LL, Shehab ZM, Wright AL, Taussig LM. Acute lower respiratory illnesses during the first three years of life: potential roles for various etiologic agents. The Group Health Medical Associates. Pediatr Infect Dis J. 1993 Jan;12(1):10-4. doi: 10.1097/00006454-199301000-00004. PMID 8380234
- [Background] Landau LI, Morgan W, McCoy KS, Taussig LM. Gender related differences in airway tone in children. Pediatr Pulmonol. 1993 Jul;16(1):31-5. doi: 10.1002/ppul.1950160107. PMID 8414738
- [Background] Duncan B, Ey J, Holberg CJ, Wright AL, Martinez FD, Taussig LM. Exclusive breast-feeding for at least 4 months protects against otitis media. Pediatrics. 1993 May;91(5):867-72. PMID 8474804
- [Background] Ray CG, Minnich LL, Holberg CJ, Shehab ZM, Wright AL, Barton LL, Taussig LM. Respiratory syncytial virus-associated lower respiratory illnesses: possible influence of other agents. The Group Health Medical Associates. Pediatr Infect Dis J. 1993 Jan;12(1):15-9. PMID 8417418
- [Background] Hampton F, Beardsmore CS, Morgan W, Williams A, Taussig L, Thompson JR. A scoring system for lung function tests in infants. Pediatr Pulmonol. 1992 Nov;14(3):149-55. doi: 10.1002/ppul.1950140303. PMID 1480440
- [Background] Wright AL, Holberg C, Martinez FD, Taussig LM. Relationship of parental smoking to wheezing and nonwheezing lower respiratory tract illnesses in infancy. Group Health Medical Associates. J Pediatr. 1991 Feb;118(2):207-14. doi: 10.1016/s0022-3476(05)80484-6. PMID 1993946
- [Background] Martinez FD, Morgan WJ, Wright AL, Holberg C, Taussig LM. Initial airway function is a risk factor for recurrent wheezing respiratory illnesses during the first three years of life. Group Health Medical Associates. Am Rev Respir Dis. 1991 Feb;143(2):312-6. doi: 10.1164/ajrccm/143.2.312. PMID 1990945
- [Background] Witt-Enderby PA, Yamamura HI, Halonen M, Palmer JD, Bloom JW. Chronic exposure to a beta 2-adrenoceptor agonist increases the airway response to methacholine. Eur J Pharmacol. 1993 Sep 7;241(1):121-3. doi: 10.1016/0014-2999(93)90942-b. PMID 7901034
- [Background] Sherrill DL, Enright PL, Kaltenborn WT, Lebowitz MD. Predictors of longitudinal change in diffusing capacity over 8 years. Am J Respir Crit Care Med. 1999 Dec;160(6):1883-7. doi: 10.1164/ajrccm.160.6.9812072. PMID 10588601
- [Background] Sherrill DL, Stein R, Halonen M, Holberg CJ, Wright A, Martinez FD. Total serum IgE and its association with asthma symptoms and allergic sensitization among children. J Allergy Clin Immunol. 1999 Jul;104(1):28-36. doi: 10.1016/s0091-6749(99)70110-7. PMID 10400836
- [Background] Sherrill D, Stein R, Kurzius-Spencer M, Martinez F. On early sensitization to allergens and development of respiratory symptoms. Clin Exp Allergy. 1999 Jul;29(7):905-11. doi: 10.1046/j.1365-2222.1999.00631.x. PMID 10383590
- [Background] Stein RT, Holberg CJ, Sherrill D, Wright AL, Morgan WJ, Taussig L, Martinez FD. Influence of parental smoking on respiratory symptoms during the first decade of life: the Tucson Children's Respiratory Study. Am J Epidemiol. 1999 Jun 1;149(11):1030-7. doi: 10.1093/oxfordjournals.aje.a009748. PMID 10355379
- [Background] Castro-Rodriguez JA, Holberg CJ, Wright AL, Halonen M, Taussig LM, Morgan WJ, Martinez FD. Association of radiologically ascertained pneumonia before age 3 yr with asthmalike symptoms and pulmonary function during childhood: a prospective study. Am J Respir Crit Care Med. 1999 Jun;159(6):1891-7. doi: 10.1164/ajrccm.159.6.9811035. PMID 10351936
- [Background] Martinez FD, Stern DA, Wright AL, Taussig LM, Halonen M. Differential immune responses to acute lower respiratory illness in early life and subsequent development of persistent wheezing and asthma. J Allergy Clin Immunol. 1998 Dec;102(6 Pt 1):915-20. doi: 10.1016/s0091-6749(98)70328-8. PMID 9847431
- [Background] Holberg CJ, Morgan WJ, Wright AL, Martinez FD. Differences in familial segregation of FEV1 between asthmatic and nonasthmatic families. Role of a maternal component. Am J Respir Crit Care Med. 1998 Jul;158(1):162-9. doi: 10.1164/ajrccm.158.1.9706117. PMID 9655724
- [Background] Lebowitz MD, Sherrill DL, Kaltenborn W, Burrows B. Peak expiratory flow from maximum expiratory flow volume curves in a community population: cross-sectional and longitudinal analyses. Eur Respir J Suppl. 1997 Feb;24:29S-38S. PMID 9098707
- [Background] Lebowitz MD. Age, period, and cohort effects. Influences on differences between cross-sectional and longitudinal pulmonary function results. Am J Respir Crit Care Med. 1996 Dec;154(6 Pt 2):S273-7. doi: 10.1164/ajrccm/154.6_Pt_2.S273. No abstract available. PMID 8970400
- [Background] Sherrill D, Viegi G. On modeling longitudinal pulmonary function data. Am J Respir Crit Care Med. 1996 Dec;154(6 Pt 2):S217-22. doi: 10.1164/ajrccm/154.6_Pt_2.S217. PMID 8970391
- [Background] Lombardi E, Stein RT, Wright AL, Morgan WJ, Martinez FD. The relation between physician-diagnosed sinusitis, asthma, and skin test reactivity to allergens in 8-year-old children. Pediatr Pulmonol. 1996 Sep;22(3):141-6. doi: 10.1002/(SICI)1099-0496(199609)22:33.0.CO;2-S. PMID 8893251
- [Background] Lebowitz MD. Epidemiological studies of the respiratory effects of air pollution. Eur Respir J. 1996 May;9(5):1029-54. doi: 10.1183/09031936.96.09051029. PMID 8793468
- [Background] Wright AL, Holberg CJ, Morgan WJ, Taussig LM, Halonen M, Martinez FD. Recurrent cough in childhood and its relation to asthma. Am J Respir Crit Care Med. 1996 Apr;153(4 Pt 1):1259-65. doi: 10.1164/ajrccm.153.4.8616551.
- [Background] Habib MP, Burrows B : Chronic Airways Obstruction: The Importance of Certain Risk Factors for Its Development. In: Current Pulmonology. DH Simmons (Ed), Year Book Medical Publishers, 1989.
- [Background] Martinez FD. Viral infections and the development of asthma. Am J Respir Crit Care Med. 1995 May;151(5):1644-7; discussion 1647-8. doi: 10.1164/ajrccm/151.5_Pt_1.1644. PMID 7735627